CLINICAL TRIAL: NCT00543972
Title: An Open Label, Dose-Escalation Safety and Pharmacokinetic Study of AVE9633 Administered as a Single Agent by Intravenous Infusion on Day 1, Day 4 and Day 7 of a 4-Week Cycle in Patients With Relapsed or Refractory CD33-Positive Acute Myeloid Leukemia (AML)
Brief Title: Dose Escalation Safety and Pharmacokinetic Study of AVE9633 as Single Agent in Relapsed/Refractory CD33-Positive Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: due to absence of evidence of clinical activity up to toxic doses
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED10219; EudraCT 2006-005976-41
Record Dates: First submitted 2007-10-12; First posted 2007-10-15 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-05

CONDITIONS: Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid | interventions — AVE9633

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AVE9633 — Intravenous Infusion

SUMMARY:
The primary objective is to determine the maximum tolerated dose of AVE9633 and to characterize the dose limiting toxicity(ies). Secondary objectives are to determine the anti-leukemia activity, the global safety and the PK profile.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CD33-positive acute myeloid leukemia, refractory or relapsed after standard treatment with no curative option available
* ECOG performance status 0 to 2

Exclusion Criteria:

* Therapy with gemtuzumab ozogamicin (Mylotarg) within 6 months prior to inclusion
* Allogenic transplantation within 6 months prior to inclusion
* Prior therapy (chemotherapy, targeted agents, radiotherapy) within 3 weeks except for hydroxyurea and for leukophoresis
* Previous treatment with AVE9633
* Poor kidney, liver and bone marrow functions
* Any serious active disease or co-morbid condition, which in the opinion of the principle investigator, will interfere with the safety or with compliance with the study
* Pregnant or breast-feeding women
* Patient with reproductive potential without effective birth control methods

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicity(ies) at each tested dose level | Study period

SECONDARY OUTCOMES:
Complete Remission (CR) / Remission with incomplete platelet recovery (CRp), Partial Remission (PR) rate, time to CR and duration of CR, peripheral blast clearance | Study period
Incidence of Adverse Events | Study period

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (3):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Barcelona, Spain